CLINICAL TRIAL: NCT05779956
Title: Personalized Medicine for Spinal Muscular Atrophy: a Translational Project to Achieve Patient Specific Therapeutic Guidance.
Brief Title: Personalized Medicine for SMA: a Translational Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Milan (Other); Ospedale Pediatrico Bambino Gesu (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3730
Record Dates: First submitted 2023-02-27; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: biomarkers,; spional muscular atrophy;; outcome
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major breakthroughs in the treatment for Spinal muscular atrophy (SMA) have been recently achieved with various therapeutic approaches that increase full-length SMN protein levels. The variability observed following the advent of commercial availability of Nusinersen for all types of SMA has highlighted the need to identify tools that may allow to predict possible therapeutic responses. The aim of this project is to establish whether an integrated approach using clinical, imaging (muscle MRI) and circulating biomarkers, can provide the possibility to develop a predictive model of therapeutic response to novel therapies for SMA patients. More specifically we wish to establish the correlation between clinical response, different biomarkers indicative of central nervous system efficacy (e.g. determination of neurofilaments levels), and markers that provide evidence of the skeletal muscle response (e.g. serum myostatin and muscle imaging) in different types of SMA

DETAILED DESCRIPTION:
Hyphotesis and Significance:

The individual variability in clinical response to treatment reported in the first Nusinersen studies has been confirmed by post approval real-world data. While some children acquire unexpected motor abilities, others have an apparently more limited clinical response. Age at disease onset and severity are reported to play a role, but do not account for the entire spectrum of clinical responses observed. There is a strong need to identify clinical and laboratory biomarkers to better understand the variables that determine the response to treatment in individuals, especially under the prospect of having further therapeutic options approved in the near future.

Working hypothesis: The hypothesis is that circulating, including neurofilaments and myostatin pathway, and imaging biomarkers may provide additional information to clinical longitudinal data and that an integrated approach may provide a better possibility to develop a predictive model of therapeutic response to novel therapies for SMA patients.

The aim is to to set up a platform of biomarkers, including circulating NfL, myostatin pathway (GDF8, FOLLISTATIN, GDF11 and ACTIVIN A) and creatinine, to establish how they relate to clinical findings and to better understand if these variables may determine clinical response to the treatment in SMA.

In patients older than 5 years, muscle MRI at baseline will also be used to explore if the pattern and severity of muscle involvement can better define the phenotype and predict therapeutic response

Specific Aim 2:

to identify trajectories of clinical progression in patients treated with Nusinersen, using our prospective data in combination with available data in other patients recently treated with Nusinersen

Specific Aim 3:

The overarching aim of this project is to explore the possibility to develop an integrated predictive model of therapeutic response to novel therapies for SMA patients

ELIGIBILITY:
Inclusion Criteria:

* All patients with SMA undergoing one of the treatments provided as standards of care

Exclusion Criteria:

* untreated patients
* patients/crarers unwilling to sign consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all pèatients withj a genetically confirmed diagnosis of 5Q spinal muscular atrophy who receive a treatment as part of standards of care
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
neurofilament levels | 3 years
  serum and CSF neurofilament levels to be determined n relation to age and severity
miostatin levels | 3 years
  Serum levels to be determined in relation to age and severity
Hammesrmith Functional motor Scale expanded | 3 years
  motor functional scale, minimum score 0, maximum score 74 indicating best performance

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, MD, Principal Investigator — F Policlinico Gemelli IRCCS
Locations (2):
- Italy (2):
  - Ospedale Bambino gesu, Rome
  - Policlinico gemelli, Rome

IPD SHARING:
Plan to Share IPD: No
aggregate data only in line with italian regulation and consnet